CLINICAL TRIAL: NCT04887714
Title: Physiological Impact of Cloth Mask During Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MaskStudy
Record Dates: First submitted 2021-05-01; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mask (Experimental): cloth mask wearing
  Interventions: Other: Mask
- control (No Intervention): control, without mask.

INTERVENTIONS:
Other: Mask — Mask wearing
  Arms: Mask

SUMMARY:
Mask wearing during the Covid-19 pandemic has been proven substantially effective in containing the spread of infection, with cloth masks being the most universally used. However, cloth masks may be uncomfortable and have physiological repercussion during exercise. This study aims to investigate the impact of cloth masks during exercise.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* active, non-active and athletic individuals;

Exclusion Criteria:

* preexisting chronic conditions
* obesity
* physical limitation precluding exercise.

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-05-07 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
perceived exertion ratings | immediately after the intervention
  assessed by a scale (7 to 20, with higher values meaning higher perceived exertion)
perceived exertion ratings | during the intervention
  assessed by a scale (7 to 20, with higher values meaning higher perceived exertion)

SECONDARY OUTCOMES:
oxygen consumption | immediately after the intervention
  assessed by cardiopulmonary test
spirometry/lung function (VeVCO2 Slope) | during the intervention
  assessed by cardiopulmonary test
spirometry/lung function (PetCO2) | during the intervention
  assessed by cardiopulmonary test
spirometry/lung function (OUES) | during the intervention
  assessed by cardiopulmonary test
spirometry/lung function (flow-volume loop) | during the intervention
  assessed by cardiopulmonary test
blood lactate | immediately after the intervention
  assessed by lactate analyzer
oxygen saturation | immediately after the intervention
  assessed by pulse oximetry
vertical jump | immediately after the intervention
  assessed by jump test
heart rate recovery | immediately after the intervention
  assessed by heart rate monitor
Scale of Measuring Subjective Perceptions to maskwearing | immediately after the intervention
  assessed by a scale (0 to 10, with higher values meaning more uncomfortable)

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital - School of Medicine - University of Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD will be make available upon reasonable request.

REFERENCES:
- [Derived] Marticorena FM, Barreto GC, Guardieiro NM, Esteves GP, Oliveira TN, de Oliveira LF, Pinto ALS, Riani L, Prado DM, Saunders B, Gualano B. Performing moderate to severe activity is safe and tolerable for healthy youth while wearing a cloth facemask. PLoS One. 2023 Mar 6;18(3):e0282475. doi: 10.1371/journal.pone.0282475. eCollection 2023. PMID 36877666
- [Derived] Guardieiro NM, Barreto G, Marticorena FM, Nunes Oliveira T, de Oliveira LF, Pinto ALS, Prado DMLD, Saunders B, Gualano B. A Cloth Facemask Causes No Major Respiratory or Cardiovascular Perturbations During Moderate to Heavy Exercise. J Phys Act Health. 2022 Dec 7;20(1):35-44. doi: 10.1123/jpah.2022-0145. Print 2023 Jan 1. PMID 36476970